CLINICAL TRIAL: NCT05570825
Title: A Phase 2 Trial of SX-682 and Pembrolizumab in Patients With Treatment Naive Stage IV or Recurrent Non-Small Cell Lung Cancer
Brief Title: SX-682 With Pembrolizumab for the Treatment of Metastatic or Recurrent Stage IIIC or IV Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Syntrix Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1122737; NCI-2022-07428 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P50CA228944 (NIH); 11019 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SX-682, pembrolizumab) (Experimental): Patients receive SX-682 PO BID, starting 7 days prior to the start of pembrolizumab, and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy and PET/CT or CT at screening and on study and undergo MRI and collection of blood samples at screening, throughout the study, and during follow up.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: CXCR1/2 Inhibitor SX-682; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: CXCR1/2 Inhibitor SX-682 — Given PO
  Other Names: SX 682; SX-682; SX682
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475; BCD-201; Pembrolizumab Biosimilar BCD-201; GME 751
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial tests whether CXCR1/2 inhibitor SX-682 (SX-682) with pembrolizumab works to treat patients with stage IIIC or IV non-small cell lung cancer that has spread to other parts of the body (metastatic) or that has come back (recurrent). SX-682 is a drug that binds to receptors on some types of immune and cancer cells, inhibiting signaling pathways, reducing inflammation, and allowing other types of immune cells to kill and eliminate cancer cells. Pembrolizumab is a monoclonal antibody that binds to a receptor called PD-1 that is found on the surface of T-cells (a type of immune cell), activating an immune response against tumor cells. Giving SX-682 in combination with pembrolizumab may be more effective at treating patients with metastatic or recurrent non-small cell lung cancer than giving these treatments alone.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive SX-682 orally (PO) twice daily (BID), starting 7 days prior to the start of pembrolizumab, and pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy and positron emission tomography (PET)/computed tomography (CT) or CT at screening and on study and undergo magnetic resonance imaging (MRI) and collection of blood samples at screening, throughout the study, and during follow up.

After completion of study treatment, patients are followed up for up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years and older
* Pathologically or cytologically confirmed non-small cell lung cancer with no known oncogenic EGFR mutation, ALK rearrangement, ROS1 rearrangement or RET rearrangement
* Tumoral PD-L1 expression >=1% by any Clinical Laboratory Improvement Act (CLIA)-certified assay
* Metastatic or recurrent non-small cell lung cancer (NSCLC). Stage IIIC per 8th edition TNM stage classification is allowed if not amenable to curative surgery or radiation per investigator judgment
* At least one site of measurable disease as determined by the Investigator, using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1. Subjects must have ECOG PS 0 or 1 at the time of informed consent and at the time of treatment initiation
* Must be willing to provide pre-treatment archived specimen or undergo a biopsy procedure if archived specimen is not available
* Must be willing to provide an on-treatment biopsy, if deemed safe by the treating physician
* Platelet count >= 100,000/uL
* Absolute neutrophil count >= 1,500/uL
* Hemoglobin >= 8g/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times upper limit of normal
* Creatinine =< 2.0 mg/dL
* Women of child-bearing potential and sexually active men must agree to use adequate contraception (hormonal or barrier method) prior to treatment initiation, during treatment and for three months after completing treatment
* Negative beta-human chorionic gonadotropin (hCG) pregnancy test at screening for patients of childbearing potential. Pregnant or breast feeding women are not eligible
* Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

* Participants must not have received prior chemotherapy or immune checkpoint inhibitor or immune-modulatory therapy (e.g. anti-PD[L]1, anti-CTLA4, anti-TIM3, anti-GITR, anti-TIGIT, anti-LAG3), for metastatic or recurrent NSCLC, with the following exceptions:

  * Participants may have received prior chemotherapy, immune checkpoint inhibitor, and/or immune modulatory therapy in the curative setting if the last dose of treatment was more than (>) 24 weeks prior to consenting
  * For patients with NSCLC harboring an oncogenic alteration other than listed may have received prior small molecule inhibitor therapy (e.g. MET inhibitor for MET exon 14 mutated NSCLC). A wash-out period of at least 5 half-lives is required prior to start of study treatment
* Presence of other active cancers within the last 2 years. Patients with any prior early stage cancer who have received definitive local treatment at least 2 years previously and no evidence of recurrence are eligible. All patients with previously treated in situ carcinoma are eligible, as patients with history of non-melanoma skin cancer
* Symptomatic central nervous system (CNS) metastases; participants with known brain metastasis must be asymptomatic with no steroids or escalating doses of antiepileptics within 7 days prior to start of study treatment

  * Patients with untreated CNS metastases may be enrolled as long as they meet the above criteria. Patients with bulky CNS metastases should consider receiving radiation prior to study entry per investigator judgment
* Participants with spinal cord compression must have received local treatment and must have been symptomatically stable with no use of steroids for at least 7 days prior to start of study treatment
* Participants must not have an active autoimmune disease that has required immune modulating treatment within (<) 365 days prior to consenting (i.e., disease modifying agents, corticosteroids). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed
* Inability to discontinue systemic corticosteroid therapy; systemic steroids must be tapered off 7 days prior to first dose of SX-682
* Known history of primary immunodeficiency
* History of organ transplant that requires use of immunosuppressives
* Current symptomatic pneumonitis and any past history of immune checkpoint inhibitor related pneumonitis regardless of steroid treatment history
* History of non-infectious pneumonitis (e.g. radiation pneumonitis) that required steroids within 3 months of start of study treatment
* Radiotherapy within 7 days of start of study treatment
* Major surgery within 21 days of start of study treatment. Minor surgery within 2 weeks of start of study treatment. Placement of vascular access device and biopsies are not considered major or minor surgery and are allowed
* Electrocardiogram (EKG) demonstrating a corrected QT (QTc) interval > 480 msec on three consecutive EKGs or patients with congenital long QT syndrome
* Severe lung disease (e.g. chronic obstructive pulmonary disease [COPD]) who cannot stop steroids 7 days prior to start of study treatment
* Serious cerebrovascular and cardiac disease defined as:

  * Active unstable angina pectoris
  * Congestive heart failure NYHA (New York Heart Association) > grade 3
  * Acute myocardial infarction within 3 months of consenting
  * Stroke or transient ischemic attack within 3 months of consenting
* Known active chronic infections: Active hepatitis B, hepatitis C and tuberculosis. Testing is not required for assessment of eligibility. Active infection requiring IV antibiotics within 7 days of study treatment initiation

  * Hepatitis C virus (HCV) infection: Patients with known history of HCV infection are eligible if HCV viral load is below the limit of quantification per local assay
  * Hepatitis B virus (HBV) infection: Patients with known history of HBV infection are eligible if HBV viral load is below the limit of quantification and negative hepatitis B virus surface antigen (HBsAg) per local assay
* Known uncontrolled HIV (human immunodeficiency virus) infection

  * Participants with known HIV infection are allowed if they are receiving anti-retroviral therapy, have CD4+ T-cell count >= 350 cells/uL within 6 months prior to study treatment initiation and no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection
* Any serious or uncontrolled concomitant disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Best objective response rate | Up to 6 years
  Response is defined as a complete response (CR) or partial response (PR) as best objective response.
  For the primary analyses, binary proportions will be estimated along with 90% confidence intervals (consistent with 1-sided 5% level testing).

SECONDARY OUTCOMES:
Response rate within subgroups | Up to 6 years
  Will be defined by low and high tumor proportion score (TPS) separately (if there are sufficient numbers of low TPS, will evaluate the high TPS group). The response rates and associated 80% confidence intervals will be estimated.
Disease control rate | Up to 6 years
  Will be defined as CR, PR, or stable disease.
Duration of response | Date of first documentation of confirmed response (CR or PR) to date of first documentation of progression, assessed up to 6 years
  Will be estimated using the method of Kaplan-Meier. Confidence intervals about medians will be estimated using the Brookmeyer-Crowley method.
Progression-free survival | Date of study registration to date of first documentation of progression, assessed up to 6 years
  Will be estimated using the method of Kaplan-Meier. Confidence intervals about medians will be estimated using the Brookmeyer-Crowley method.
Overall survival | Date of study registration to date of death due to any cause, assessed up to 6 years
  Will be estimated using the method of Kaplan-Meier. Confidence intervals about medians will be estimated using the Brookmeyer-Crowley method.
Frequency and severity of adverse events | Up to 6 years
  Toxicity frequencies will be estimated with 95% confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Christina S. Baik, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No